CLINICAL TRIAL: NCT06694207
Title: Effect of Intraperitoneal Bupivacaine with Dexmedotomidine or Fentanyl for Post-Operative Analgesia Following Laparoscopy in Pediatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Youssef Roshdy Kelada, Wessam Nashaat Ali Mohamed, Assiut University
Other Study IDs: Intraperitoneal Bupivacaine
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Post Operative Analgesia
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Intraperitoneal Bupivacaine with Dexmedotomidine or Fentanyl — Intraperitoneal Bupivacaine with Dexmedotomidine or Fentanyl for Post-Operative Analgesia Following Laparoscopy in Pediatric Patients

SUMMARY:
To compare analgesic effect of adding dexmedomedin or fentanyl to intraperitoneal bupivacain in pediatric patients undergoing laparoscopy. The primary outcome is to compare pain using the Children's Hospital of Eastern Ontario score (CHEOPS). The secondary goal is to compare the time to the first request for analgesia in the post-operative period, the total dose of analgesics used in the 24 hours (post-operative), side effects, and signs of systemic absorption and toxicity.

DETAILED DESCRIPTION:
Laparoscopic procedures have many advantages over open procedures such as lesser hemorrhage , better cosmetic results, lesser postoperative pain and shorter recovery time leading to a shorter hospital stay and less expenditure . Laparoscopic procedures are associated with postoperative pain affecting early ambulation of the patient. Pain in laparoscopic surgery results from stretching of the abdominal cavity, peritoneal inflammation, diaphragmatic irritation and residual carbon dioxide (CO2) in the peritoneal cavity . Peritoneal irritation by carbonic acid (formed by reaction between carbon dioxide CO2 and water) and the creation of space between the liver and diaphragm by residual pneumoperitoneum has been implicated for visceral and shoulder tip pain. Humidity and volume of the insufflated gas, wound size, and trauma to the parietal peritoneum may also be responsible for this pain. A multimodal approach is required to alleviate all three types of pain which includes parenteral NSAIDs, opioids, and postoperative intraperitoneal local anesthetic instillation, port-site infiltration of local anesthetic, intra-peritoneal saline, removal of insufflation gas, gas drains, low-pressure abdominal insufflations, acetazolamide administration and use of N2O in place of CO2, etc. Intraperitoneal local anesthetic (IPLA) appears promising in pediatric surgery although the high absorptive capacity of the peritoneum and high peritoneal surface area in children. Hence, the delivery of an effective dose without toxicity in children could be challenging. Fentanyl selectively binds to the mu-receptor in the central nervous system (CNS). Stimulation of the mu-subtype opioid receptor stimulates the exchange of GTP for GDP on the G-protein complex and subsequently inhibits adenylate cyclase, so decreasing in intracellular cAMP and leads to a reduction in the release of neurotransmitters. It was found that administering either fentanyl or ketamine as an LA adjuvant dramatically speed up the onset of anesthesia, prolonged the duration of lid akinesia, increased the duration of globe akinesia, and lengthened the time for the first request of postoperative analgesia. Opioids, in conjunction with local anesthetics, improve the quality of intraoperative analgesia and prolong the duration of postoperative analgesia. Although morphine was the first opioid used, a wide variety of clinically relevant side effects, especially respiratory depression, limited its utility. In contrast, a favorable pharmacokinetic and pharmacodynamic profile of lipophilic opiates (fentanyl) proved to be a better alternative as their lipophilicity leads to rapid uptake and faster clinical onset of action and short duration of action. Dexmedetomidine (alpha-2 adrenergic agonists) has become one of the frequently used drugs in anesthesia as it has been reported to provide analgesia, anxiolysis, and an anesthetic-sparing action with minimal respiratory depression plus its sedative effect that mimics natural sleep. Intraperitoneal instillation of dexmedetomidine with bupivacaine reduces the pain after elective laparoscopy in adults as compared to that with bupivacaine alone or with tramadol. In addition, the postoperative requirement for rescue analgesia is reduced. The purpose of the study is to assess and compare the analgesic effectiveness of intraperitoneal bupivacaine in paediatric patients with either fentanyl or Dexmedotomidine.

ELIGIBILITY:
Inclusion Criteria:

Who will undergo laparoscopy.

Exclusion Criteria:

Children with a known history of Heart disease, Local anesthetic allergy, and Body mass index of ≥95th percentile for age.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This prospective study will include pediatric patients who will be admitted to hospitals of Assuit University including Children from both sexes, Children aged 6-9 years old, Have the American Society of Anesthesiologists (ASA) physical status I or II and those who will undergo laparoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to compare pain using the Children's Hospital of Eastern Ontario score (CHEOPS) | Baseline
  compare the time to the first request for analgesia in the post-operative period, the total dose of analgesics used in the 24 hours (post-operative), side effects, and signs of systemic absorption and toxicity

REFERENCES:
- [Background] Kaarthika T, Radhapuram SD, Samantaray A, Pasupuleti H, Hanumantha Rao M, Bharatram R. Comparison of effect of intraperitoneal instillation of additional dexmedetomidine or clonidine along with bupivacaine for post-operative analgesia following laparoscopic cholecystectomy. Indian J Anaesth. 2021 Jul;65(7):533-538. doi: 10.4103/ija.IJA_231_21. Epub 2021 Jul 23. PMID 34321684